CLINICAL TRIAL: NCT06218082
Title: Vitiligo Registry for Adults and Children in the UK (VIRTUAL-UK)
Brief Title: Vitiligo Registry for Adults and Children in the UK
Acronym: VIRTUAL-UK
Status: Not yet recruiting | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Collaborators: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022DER127
Record Dates: First submitted 2022-11-15; First posted 2024-01-23 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Dermatologic Disease; Vitiligo
MeSH Terms: conditions — Skin Diseases; Vitiligo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vitiligo is the most common depigmentation disorder affecting around 1% of the population worldwide. Fifty two percent of patients develop vitiligo before the age of 20 and around 80% develop vitiligo before the age of 30 years old.1 Vitiligo often presents in childhood and tends to be a lifelong disease, requiring prolonged courses of phototherapy.

Currently no national or international registry for patients with vitiligo exists. Individual dermatologists maintain a database of such patients, however no coordinated efforts have been made to combine these individual registries into a broader national registry. Finally, recently published British Association of Dermatologists (BAD) guideline for the management of vitiligo, recommended the development of a national registry for people with vitiligo undergoing systemic or light therapy to identify outcomes and safety.

DETAILED DESCRIPTION:
Vitiligo is the most common depigmentation disorder affecting around 1% of the population worldwide. Fifty two percent of patients develop vitiligo before the age of 20 and around 80% develop vitiligo before the age of 30 years old. Vitiligo often presents in childhood and tends to be a lifelong disease, requiring prolonged courses of phototherapy.

Vitiligo is an autoimmune skin disorder and is often associated with multiple other autoimmune disorders such as thyroid disorders, diabetes, IBS, pernicious anemia, alopecia areata amongst others. Current treatments include topical corticosteroids and calcineurin inhibitors, phototherapy, combination of phototherapy with oral corticosteroids, laser and surgical interventions. Other treatment modalities such as Methotrexate have also been trialed. Currently available treatments are being used off license with uncertain therapeutic success.

Previously, it has been shown that vitiligo has an inverse relationship with melanoma, which means that people with vitiligo are less likely to develop melanoma. A recent systematic review and meta-analysis looking into the risk of skin cancer in people with vitiligo showed that compared with people without vitiligo, people with vitiligo had a significantly lower risk of nonmelanoma skin cancer. The same pattern occurred for melanoma (but was not statistically significant). However, this review was limited by the small number of included studies and high heterogeneity due to methodological and clinical differences between the included studies. In addition, there is lack of data on the skin cancer risk for vitiligo patients who receive prolonged phototherapy courses, especially regarding high cumulative exposures in children with less deeply pigmented skin. This is especially important when NB-UVB is combined with topical tacrolimus treatment, due to theoretical increased risk of skin cancer.

In addition, there is an urgent need for new, effective and licensed treatment for vitiligo. In the dawn on new therapeutic era of new emerging treatments such as topical and oral JAK inhibitors, evidence will be needed on the effectiveness, safety and cost effectiveness of such therapies compared to other treatments. In order to gather evidence on clinical effectiveness of vitiligo treatments and to assist with updating of clinical guidance pathway, as well as to gather information on possible risk factors, adverse events, maintenance regime and assist with conduction of post marketing studies, prospective multicentre registry is needed for vitiligo patients who are treated with phototherapy, combination treatments (with phototherapy), oral agents (such as oral corticosteroids) including new emerging JAK inhibitors (once there are available in the UK).

Oral corticosteroids combined with phototherapy are recommended by the recently published BAD guidelines for cases of rapidly progressive vitiligo. Case reports were published on initiation of methotrexate and oral JAK inhibitors for the treatment of vitiligo.

In addition, there is no firm data on disease progression and especially predictors of rapidly progressive vitiligo are largely unknown, which is a challenging scenario for the patient and their clinician.

Currently no national or international registry for patients with vitiligo exists. Individual dermatologists maintain a database of such patients, however no coordinated efforts have been made to combine these individual registries into a broader national registry. Finally, recently published British Association of Dermatologists (BAD) guideline for the management of vitiligo, recommended the development of a national registry for people with vitiligo undergoing systemic or light therapy to identify outcomes and safety.2

As an initial, preliminary step for the development of the online UK registry for vitiligo patients, development of a pilot multi-centred registry in the UK is needed. In addition, such registry will be co-ordinated with a pilot multi-centred registry in France and the USA. Each registry will be developed separately (country-specific) and there will be no data sharing between the registries, however there will be co-ordination between the CIs of the registries with regards to the outcomes collected.

Another challenge in vitiligo has been consistency in the use of core outcome domains and measures instruments to define treatment success or failure. The international Initiative for Outcomes for vitiligo (INFO) has previously addressed this heterogeneity and defined 3 outcome domains as being essential: repigmentation, side effects/harms and maintenance of gained repigmentation. Four items were further recommended for inclusion but were not considered to be essential: cosmetic acceptability of the results, quality of life, cessation of spreading of vitiligo and tolerability or burden of treatment.5 INFO has subsequently published recommendations on how to measure repigmentation in target lesion. Percentage of repigmentation in quartiles (0-25%, 26-50%, 51-79%, 80-100%) should be measured as well as cosmetic acceptability of results should be assessed using the Vitiligo Noticeability Scale.6 There are also several other established instruments exist (such as VASI, VIPs, VITs) to measure these domains and these are suitable for use in a registry.

A long-term safety data will be vital to provide pharmacovigilance, particularly regarding rare or delayed adverse effects of treatment. Hence a prospective multicentre registry study is greatly needed to evaluate the real-world use of phototherapy (including combination treatments with phototherapy), topical JAK inhibitors, systemic immuno-modulatory therapies in adults and children undergoing treatment for vitiligo to provide effectiveness and safety data beyond the confines of short-term randomised controlled trials (RCTs). Such a registry will ultimately inform treatment guidelines, provide pharmacogenetic and pharmacodynamic research data, and help to identify those patients likely to experience rapid disease progression, ultimately improving and personalising patient care. With novel topical and oral immunomodulatory therapies having just entering vitiligo clinical practice, the timing is ideal to harness the high-quality data collection offered by the UK NHS.

ELIGIBILITY:
Inclusion Criteria:

1. Paediatric and adult patients with vitiligo under management in secondary care.
2. Written informed consent for study participation obtained from the patient or parents / legal guardian, with assent as appropriate by the patient, depending on the level of understanding.
3. Participants consent to participate in long-term follow up and access to all relevant medical records as needed by the study team
4. Clinical diagnosis of vitiligo made by a dermatologist
5. Willingness to comply with all study requirements.
6. Competent use of English language, according to patient's age (capable of understanding patient questionnaires).

Exclusion Criteria:

1. Insufficient understanding of the study by the patient and/or parent/guardian.
2. Patients with vitiligo/their parents or guardians, who do not provide consent for participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients (adults and children) seen at various hospitals in the UK and who are diagnosed with vitiligo will be included. Vitiligo patients who receive therapy with systemic steroids, phototherapy including laser, surgical treatments, new immunomodulators (e.g. topical or oral JAK inhibitor) once they enter UK market and any combination therapies of the above will be eligible to be included in the registry.
  There is no upper or lower age limit for participation. The decision to therapy or switch to another systemic agent will be the result of the treating dermatology consultant's decision, following discussion with the patient/parent/legal guardian, without using a pre-specified severity score cut off. It is the treating physician's responsibility to ensure that patients are suitable for the therapy, and that any standard of care treatment or assessments are provided alongside participation in the study as per local requirements.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Multi-centred registry will be developed, with an aim to establish short- and long-term safety (pharmacovigilance) and effectiveness of vitiligo therapies | 12 months
  VIRTUAL-UK is a small registry and in collaboration with the BAD, aims to utilize and modify one of the existing platforms (software), in order to assist the end user (i.e. Dermatologists) in accessing the platform and reducing the time needed for training and data input.

SECONDARY OUTCOMES:
To document the clinical and socio-demographic characteristics, co-morbidities including cancers, previous treatments of patients included in the cohort as assessed by the case report forms (CRFs). | 12 months
  To document the clinical and socio-demographic characteristics, co-morbidities including cancers, previous treatments of patients included in the cohort as assessed by the case report forms (CRFs).
To describe the clinical and socio-demographic characteristics, co-morbidities including cancers, previous treatments of patients included in the cohort | 12 months
  To describe the clinical and socio-demographic characteristics, co-morbidities including cancers, previous treatments of patients included in the cohort
To assess short- and long-term safety (pharmacovigilance) of these therapies | 12 months
  To assess short- and long-term safety (pharmacovigilance) of these therapies
To evaluate the efficacy and safety of currently used therapies for vitiligo (including combination therapies), providing a basis for better shared decision making and guidelines. | 12 months
  To evaluate the efficacy and safety of currently used therapies for vitiligo (including combination therapies), providing a basis for better shared decision making and guidelines.
To evaluate the impact of these therapies on vitiligo patients' quality of life | 12 months
  To evaluate the impact of these therapies on vitiligo patients' quality of life
To attempt to identify risk factors associated with treatment failure | 12 months
  To attempt to identify risk factors associated with treatment failure
To document disease trajectory and its relationship to demographic, phenotypic and treatment factors | 12 months
  To document disease trajectory and its relationship to demographic, phenotypic and treatment factors
To develop predictors of rapidly progressive vitiligo | 12 months
  To develop predictors of rapidly progressive vitiligo

CONTACTS AND LOCATIONS:
Overall Officials: Viktoria Eleftheriadou, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom